CLINICAL TRIAL: NCT04743375
Title: Clinical Efficacy of Silk Sericin Dressing With Collagen for Split-thickness Skin Graft Donor Site Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Med Chula IRB 143/63
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Wound Heal; Wound Surgical; Donor Site Complication
Keywords: Wound dressing; Sericin; Collagen; Split-thickness skin graft donor site (STSG donor site)
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sericin dressing with collagen (Experimental): Sericin dressing with collagen
  Interventions: Other: wound dressing application
- Bactigras (Active Comparator): Commercial dressing
  Interventions: Other: wound dressing application

INTERVENTIONS:
Other: wound dressing application — Sericin dressing with collagen or Bactigras will be used as a primary dressing for treating the STSG donor site.

SUMMARY:
To examine the efficacy and safety of sericin dressing with collagen in STSG donor site treatment comparing with Bactigras®. Around 30 patients will be enrolled in this study.

DETAILED DESCRIPTION:
Wounds are a public health problem found worldwide that associated with both clinical and economic burdens. Although several wound dressings are available, some limitations of those dressings still existed resulting in the need for new wound dressing development.

The sericin dressing with collagen was developed to provide a moist environment and bioactive ingredients to the wound bed. To evaluate its efficacy and safety, the STSG donor sites of each patient will be divided into two equal areas. Each area will be randomly allocated into sericin dressing with collagen group or control group (Bactigras®). The outcomes will be collected to examine the efficacy and safety of sericin dressing with collagen in comparison with commercial dressing Bactigras®.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have STSG donor site wounds on the thigh area
* Age more than 18 years old
* The split-thickness skin graft is harvested for the first time at the investigated area.
* Patients who are able to communicate with the Thai language
* Willingness to participate

Exclusion Criteria:

* Patient with a mental disorder or immunocompromised diseases
* Patients who cannot or not willing to follow the protocol
* Known sensitivity or allergy to sericin, chlorhexidine, and collagen
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Time to complete healing | 42 days
  The number of days since starting treatment until the primary dressing can spontaneously detach from wound with full re-epithelialization (at least 95% re-epithelialization) without any drainage.

SECONDARY OUTCOMES:
Pain score | 42 days
  Pain score evaluated by patient using visual analog scales (0-10)
Incidence of infection | 42 days
  The incidence of infection will be reported as "present" or "not present". Infection wound is wound which has purulent secretion or some of the inflammatory reactions (erythema, warmth, pain or tenderness, or induration) and has positive result from microbiological test.
Incidence of adverse effect | 42 days
  Adverse effects on hepatic function, renal function, and other adverse effects resulted from dressing application will be reported as "present" or "not present".
Vancouver scar scale (VSS) | 6 months
  Vancouver scar scale evaluated by clinician at 1, 3, and 6 months after complete wound healing
Patient scale of Patient and observer scar scale (POSAS) | 6 months
  Patient scale of Patient and observer scar scale (POSAS) evaluated by patients 6 months after complete wound healing
Erythema level | 6 months
  Erythema level measured by using Mexameter® at 1, 3, and 6 months after complete wound healing
Melanin level | 6 months
  Melanin level measured by using Mexameter® at 1, 3, and 6 months after complete wound healing
Trans-epidermal water loss (TEWL) | 6 months
  TEWL measured by using Tewameter® at 1, 3, and 6 months after complete wound healing
Skin hydration | 6 months
  Hydration level measured by using Corneometer® at 1, 3, and 6 months after complete wound healing
Skin elasticity | 6 months
  Elasticity parameters measured by using Cutometer® at 1, 3, and 6 months after complete wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Ph.D, Principal Investigator — Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn University
Locations (1):
- Chulalongkorn Hospital, Bangkok, Thailand